CLINICAL TRIAL: NCT06259526
Title: A Phase 2, Multi-Center, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Effectiveness and Safety of JS1-1-01 in Patients With Moderate to Severe Depression
Brief Title: A Study of the Effectiveness and Safety of JS1-1-01 in Patients With Moderate to Severe Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSL-CM-JS1-1-01-Ⅱ
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo group
- JS1-1-01 low-dose group (Experimental)
  Interventions: Drug: JS1-1-01 low-dose group
- JS1-1-01 medium dose group (Experimental)
  Interventions: Drug: JS1-1-01 pills; JS1-1-01 placebo pills; Duloxetine hydrochloride placebo capsules
- JS1-1-01 high-dose group (Experimental)
  Interventions: Drug: JS1-1-01 high-dose group
- Active drug group (Active Comparator)
  Interventions: Drug: Active drug group

INTERVENTIONS:
Drug: Placebo group — (1 pill of 25 mg JS1-1-01 placebo pills +1 pill of 50 mg JS1-1-01 placebo pills+1 pill of duloxetine hydrochloride placebo capsule)/time, 2 times per day, administered postprandial, for 8 consecutive weeks.
  Other Names: JS1-1-01 placebo pills; Duloxetine hydrochloride placebo capsules
  Arms: Placebo group
Drug: JS1-1-01 low-dose group — (1 pill of 25 mg JS1-1-01 pills +1 pill of 50 mg JS1-1-01 placebo pills +1 pill of duloxetine hydrochloride placebo capsule)/time, 2 times/day, administered postprandial, for 8 consecutive weeks.
  Other Names: JS1-1-01 pills; JS1-1-01 placebo pills; Duloxetine hydrochloride placebo capsules
  Arms: JS1-1-01 low-dose group
Drug: JS1-1-01 pills; JS1-1-01 placebo pills; Duloxetine hydrochloride placebo capsules — (1 pill of 25 mg JS1-1-01 placebo pills+1 pill of 50 mg JS1-1-01 pills +1 pill of Duloxetine hydrochloride placebo capsule)/time, 2 times/day, administered postprandial, for 8 consecutive weeks.
  Other Names: JS1-1-01 pills; JS1-1-01 placebo pills
  Arms: JS1-1-01 medium dose group
Drug: JS1-1-01 high-dose group — (1 pill of 25 mg JS1-1-01 pills +1 pill of 50 mg JS1-1-01 pills +1 pill of Duloxetine hydrochloride placebo capsule)/time, 2 times per day, administered postprandial, for 8 consecutive weeks.
  Other Names: JS1-1-01 pills; Duloxetine hydrochloride placebo capsules
  Arms: JS1-1-01 high-dose group
Drug: Active drug group — (1 Duloxetine hydrochloride enteric coated capsule+1 pill of 25mg JS1-1-01 placebo pills+1 pill of 50mg JS1-1-01 placebo pills)/dose, 2 times per day, administered postprandial, for 8 consecutive weeks.
  Other Names: JS1-1-01 placebo pills; Duloxetine hydrochloride enteric coated capsule
  Arms: Active drug group

SUMMARY:
The purpose of this study is to evaluate the Effectiveness and Safety of JS1-1-01 in Patients With Moderate to Severe Depression

ELIGIBILITY:
Inclusion Criteria:

* All of the following standards must be met:

  1. Age range from 18 to 65 years old (including boundary values), both male and female;
  2. Single or recurrent episodes (296.2/296.3) that meet the diagnostic criteria for depression in DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, 5th edition);
  3. During the screening and baseline periods, the total score of the Montgomery Asperger Depression Rating Scale (MADRS) was ≥ 26 points;
  4. Screening and baseline periods, with a Clinical Global Impression Scale Disease Severity (CGI-S) score of ≥ 4 points;
  5. Voluntary participation in clinical trials, able to sign informed consent forms, and able to understand and comply with research procedures.

Exclusion Criteria:

* Those who meet any of the following criteria cannot be included in this experiment:

  1. Individuals with a history of severe drug allergies or allergies to Piper Piper (pepper plant) or Duloxetine;
  2. Those who have used at least two antidepressants in sufficient dosage and duration (treated according to the maximum dosage in the instructions for at least 4 weeks) in a single or current episode in the past but still have no effect;
  3. Those who have been ineffective in using Duloxetine in sufficient amounts during the previous treatment course;
  4. The patients of depression secondary to other mental or physical illnesses;
  5. Patients of depression with accompanying psychiatric symptoms;
  6. Significant suicidal attempt or behavior within the past year, with a score of ≥ 3 on the 10th item (suicidal ideation) of the MADRS scale;
  7. During the baseline period, those with a reduction rate of ≥ 25% in the MADRS scale score compared to the screening period;
  8. Individuals with a history of epileptic seizures (excluding convulsions caused by febrile seizures in children);
  9. Individuals who have received depression related systemic physical therapy within 3 months prior to their first administration: modified electroconvulsive therapy (MECT), transcranial magnetic stimulation (TMS), vagus nerve stimulation (VNS), deep brain stimulation (DBS), phototherapy, or systemic psychotherapy;
  10. Systematically receiving antidepressant treatment within the first 2 weeks of randomization, or discontinuing antidepressant medication for less than 5 half-lives before randomization;
  11. Individuals with severe unstable cardiovascular disease, liver disease, kidney disease, blood disease, endocrine disease, and other physical diseases or medical history;
  12. Accompanied by a history of malignant tumors (excluding cured skin basal cell carcinoma and cervical carcinoma in situ);
  13. Screening or baseline electrocardiogram abnormalities that have clinical significance and are deemed unsuitable for inclusion by investigators, such as male QTcF ≥ 450 ms, female QTcF ≥ 470 ms, or having a history of long QT syndrome;
  14. A history of symptomatic orthostatic hypotension (i.e. orthostatic syncope) with clinical significance;
  15. During the screening or baseline period, TBIL is above 2 times the upper limit of normal value, and ALT or AST is above 2 times the upper limit of normal value; Cr is higher than 1.2 times the upper limit of normal value;
  16. Thyroid dysfunction (TSH above 1.2 times the upper limit of normal value or below 0.8 times the lower limit of normal value) or the presence of hyperthyroidism or hypothyroidism determined by the investigators;
  17. Individuals with a history of elevated intraocular pressure or narrow angle glaucoma;
  18. Screening period, drug abuse screening positive individuals;
  19. A history of alcohol dependence within one year prior to screening;
  20. Pregnant and lactating women, male or female subjects who have a family planning or are unable to take effective contraceptive measures within 30 days after signing the informed consent form and ending the trial;
  21. Screening for individuals who have participated in clinical trials and taken investigational drugs within the first 30 days;
  22. The investigators believe that the subjects have poor compliance or there are other clinical, social, or family factors that are not suitable for enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2023-12-26 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
The change in MADRS total score from baseline | 8 weeks
  There are a total of 10 projects in Montgomery-Asberg Depression Rating Scale（MADRS）, each with a 7-point scoring system ranging from 0 to 6 points. The higher the score, the more severe the degree of depression.

SECONDARY OUTCOMES:
The change in HAMD-17 total score from baseline | 8 weeks
  There are a total of 17 projects in Hamilton Depression Scale-17（HAMD-17）. Scores are distributed on a scale of 0 to 53. A score above 24 indicates severe depression, a score of 17 indicates moderate depression, and a score below 7 indicates no depressive symptoms.
The effective rate of MADRS | 8 weeks
  The effective definition of MADRS is that the reduction rate of MADRS score relative to baseline is ≥ 50%.
The effective rate of HAMD-17 | 8 weeks
  The effective definition of HAMD-17 is that the reduction rate of HAMD-17 score relative to baseline is ≥ 50%.
The response rate of MADRS | 8 weeks
  The response definition of MADRS is that the score ≤ 12 points.
The response rate of HAMD-17 | 8 weeks
  The response definition of HAMD-17 is that the score ≤ 7 points.
The change in CGI-I and CGI-S total score from baseline | 8 weeks
  Perform the Clinical Global Impression Scale (CGI-S) score from Visit 1 to Visit 7, and perform the Clinical Global Impression Scale (CGI-I) score from Visit 3 to Visit 7.The highest score is 7 points, and the higher the score, the more severe the condition will be.
The change in HAMA total score from baseline | 8 weeks
  There are a total of 14 projects in Hamilton Anxiety Scale（HAMA）, each with a 5-point scoring system ranging from 0 to 4 points. A total score of less than 6 on the scale is considered normal, a score of 7-14 indicates possible anxiety, a score of 15-20 indicates certain anxiety, a score of 21-28 indicates obvious anxiety, and a total score of more than 28 indicates severe anxiety. The higher the score, the more severe the anxiety.
The change in MADRS Single item score from baseline | 8 weeks
  The higher the score, the more severe the degree of depression.
The change in HAMD-17 factor score from baseline | 8 weeks
  The higher the score, the more severe the degree of depression.
The change in SHAPS total score from baseline | 8 weeks
  There are a total of 14 projects in Snaith-Hamilton Pleasure Scale（SHAPS）, each with a 4-point scoring system ranging from 1 to 4 points. Scores are distributed between 14-56 points. The higher the score, the more severe the anhedonia.

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - Capital Medical University Affiliated Anding Hospital, Beijing, Beijing Municipality
  - Peking University Sixth Hospital, Beijing, Beijing Municipality
  - Chongqing 11th People's Hospital, Chongqing, Chongqing Municipality
  - Chongqing Mental Health Center, Chongqing, Chongqing Municipality
  - The Affiliated Brain Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Hebei Provincial Mental Health Center, Baoding, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Daqing Third Hospital, Daqing, Heilongjiang
  - Wuxi Mental Health Center, Wuxi, Jiangsu
  - Zhenjiang Mental Health Center, Zhenjiang, Jiangsu
  - Jiangxi Provincial Psychiatric Hospital, Nanchang, Jiangxi
  - Jilin Provincial Neuropsychiatric Hospital, Siping, Jilin
  - Shandong Provincial Mental Health Center, Jinan, Shandong
  - Tianjin Anding Hospital, Tianjin, Tianjin Municipality
  - Ürümqi Fourth People's Hospital, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Huzhou Third People's Hospital, Huzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No